CLINICAL TRIAL: NCT01818960
Title: Revascularization Strategies for ST Elevation Myocardial Infarction; The Cardiac Magnetic Resonance Endpoint Study
Brief Title: Revascularization Strategies for STEMI; The CMR Endpoint Study
Acronym: ASSIST-CMR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC-103
Record Dates: First submitted 2013-03-23; First posted 2013-03-27 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Acute Myocardial Infarction
Keywords: Stent, Myocardial Infarction, Coronary Intervention
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SS-PCI (Active Comparator): Same sitting multivessel PCI as an adjunct to primary PCI
  Interventions: Procedure: SS-PCI
- IRA-PCI (Active Comparator): IRA only PCI with planned staging for non-IRA lesions
  Interventions: Procedure: IRA-PCI

INTERVENTIONS:
Procedure: IRA-PCI — IRA only PCI at the time of Primary PCI
  Arms: IRA-PCI
Procedure: SS-PCI — Same sitting multivessel PCI as an adjunct to primary PCI
  Arms: SS-PCI

SUMMARY:
Revascularization strategies for ST elevation myocardial infarction (STEMI) study (ASSIST-CMR) will compare the effects of two revascularization strategies [same sitting multivessel primary PCI (SS-PCI) and culprit vessel only primary PCI (IRA-PCI)] on myocardial infarct size (MIS) as determined by cardiac magnetic resonance (CMR) imaging in patients presenting with STEMI and multivessel disease (MVD).

ELIGIBILITY:
Inclusion Criteria:

* High risk ST elevation myocardial infarction evidenced by: ≥2 mm ST elevation in 2 anterior or lateral leads; or ≥2 mm ST elevation in 2 inferior coupled with ST depression in 2 contiguous anterior leads for a total ST deviation of ≥8 mm; or New left bundle branch block with at least 1 mm concordant ST elevation.
* Multivessel CAD as evidenced by ≥1 significant (≥70% by visual assessment or FFR<0.80 for 50-70% stenosis) stenosis in non-IRA.
* Successful IRA-PCI with <10% residual angiographic stenosis and TIMI III flow.
* Written informed consent.

Exclusion Criteria:

* Age ≤ 18 years.
* Prior coronary artery bypass graft (CABG) surgery.
* Administration of thrombolytic therapy.
* Non-IRA stenosis is a chronic total occlusion or located in left main artery.
* Hemodynamic instability evidenced by BP<90 mmHg, Killip class ≥2, need for inotropes/vasopressors.
* Known renal insufficiency (estimated GFR < 50ml/min).
* Contraindication to CMR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Infarct size by CMR | 90 days

SECONDARY OUTCOMES:
MACE rate | One year
  MACE rate at 12 months

OTHER OUTCOMES:
LV function | 90 days and one year

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - London Health Sciences, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Regina Qu'Appelle Health Region, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: Undecided